CLINICAL TRIAL: NCT05198544
Title: A Multi-center, Prospective Clinical Trial Evaluating a Hyaluronic Acid Matrix in the Treatment of Chronic Non-healing Diabetic Foot Ulcers (DFUs)
Brief Title: Clinical Trial Evaluating a Hyaluronic Acid Matrix in the Treatment of Chronic Non-healing Diabetic Foot Ulcers (DFUs)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SerenaGroup, Inc. (Network)
Collaborators: Lacerta Life Sciences, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACERTA-001
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: This study is a multi-center, prospective trial designed to evaluate the use of HaM in Wagner grade 1 and 2 DFUs.
  After screening, subjects are treated with weekly application of HaM and SOC for 8 weeks followed by SOC alone for the remainder of the 12-week trial period.
  The standard of care in this study consists of offloading of the DFU using a total contact cast or fixed ankle walker, sharp debridement, infection management with the use of antiseptics and proper moisture balance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hēlaquis Matrix is a hyaluronic acid matrix (HaM) (Experimental): Subjects will receive weekly application of Ham along with standard of care therapy for eight (8) weeks unless healing occurs prior to 8 weeks.
  Interventions: Device: Hēlaquis Matrix is a hyaluronic acid matrix (HaM)

INTERVENTIONS:
Device: Hēlaquis Matrix is a hyaluronic acid matrix (HaM) — Hēlaquis Matrix is a hyaluronic acid matrix (HaM) derived from the American Alligator and indicated for the treatment of chronic wounds. Hyaluronic Acid (HA) is a naturally occurring non sulphated glycosaminoglycan consisting of a linear sequence of D-glucuronic and N -acetyl-Dglucosamine. It is present in connective tissue and plays a role in several biological processes including tissue repair.

SUMMARY:
This study is a multi-center, prospective trial designed to evaluate the use of HaM in Wagner grade 1 and 2 DFUs.

After screening, subjects are treated with weekly application of HaM and SOC for 8 weeks followed by SOC alone for the remainder of the 12-week trial period.

The standard of care in this study consists of offloading of the DFU using a total contact cast or fixed ankle walker, sharp debridement, infection management with the use of antiseptics and proper moisture balance.

DETAILED DESCRIPTION:
This study is a multi-center, prospective trial designed to evaluate the use of HaM in Wagner grade 1 and 2 DFUs.

After screening, subjects are treated with weekly application of HaM and SOC for 8 weeks followed by SOC alone for the remainder of the 12-week trial period.

The standard of care in this study consists of offloading of the DFU using a total contact cast or fixed ankle walker, sharp debridement, infection management with the use of antiseptics and proper moisture balance.

The Screening Phase consists of a series of screening assessments designed to determine eligibility followed by, for those who meet the eligibility criteria, treatment.

At the Screening Visit (SV), written informed consent is obtained from the subject by the Investigator or designee prior to the performance of any other protocol-specific procedure.

At the SV, the Investigator will select the Index (study) ulcer. Each subject will have only one DFU selected as the Index (study) ulcer. If the subject has more than one ulcer at the SV, the Investigator will select the largest ulcer that meets the eligibility criteria of the protocol as the Index (study) ulcer.

The SV is designed to determine whether subjects are eligible to proceed to the Treatment Phase of the study. Those subjects who meet the eligibility criteria may transition to Treatment Visit 1 (TV1) on the same day as the SV or at a later date.

The Treatment Phase (12 Weeks) Subjects who meet eligibility criteria at the SV will receive HaM and SOC for 8 weeks followed by SOC alone for the remainder of the 12-week trial period.

During the Treatment Phase, subjects will be evaluated on a weekly basis. Efficacy evaluations each week will include Investigator assessment of ulcer healing and measurements of ulcer size using digital photographic planimetry. Safety evaluations during the Treatment Phase will consist of adverse event assessments at each visit. Subjects may receive up to eight applications of HaM. Subjects whose study ulcer does not heal after eight applications will receive only SOC treatment for 4 additional weeks. Subjects whose ulcers do not achieve closure at or by 12 weeks or who experience an amputation will be deemed treatment failures.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Presence of a diabetic foot ulcer, Wagner 1 or 2 grade, extending at least through the dermis. The ulcer may extend down to subcutaneous tissue, tendon, or muscle.
3. The ulcer must be below the medial aspect of the malleoli.
4. The index ulcer will be the largest ulcer if 2 or more ulcers are present on the same extremity. If other ulcerations are present on the same foot, they must be more than 2 cm from the index ulcer.
5. Index ulcer (i.e., current episode of ulceration) has been present for greater than 4 weeks prior to the initial screening visit.
6. Study ulcer size is a minimum of 0.75 cm2 and a maximum of 5 cm2 at first treatment visit.
7. Adequate circulation to the affected extremity as demonstrated by a transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 40 mmHg, OR an Ankle Brachial Index (ABI - measure of blood flow to the ankle) between 0.7 and 1.3 OR Toe Brachial Index greater than 0.5 within 3 months of the first Screening Visit.
8. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
9. Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
10. Subject has read and signed the IRB approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

1. Study ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
2. Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
3. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
4. History of radiation at the ulcer site.
5. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
6. Known Osteomyelitis or bone infection of the affected foot or leg as verified by diagnostic imaging within 30 days prior to enrollment.
7. Subject is pregnant or breast feeding.
8. Study ulcer with a history of treatment with hyperbaric oxygen or a cellular or Tissue-based Product (CTP) within 30 days of enrollment.
9. Subject has a known or suspected allergy to the test material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate Wound healing in Wagner 1 and 2 grade DFUs by wound size | 12 weeks
  To evaluate the effectiveness of HaM as an adjunctive treatment in facilitating complete wound healing in Wagner 1 and 2 grade DFUs when compared to well-established standard of care healing rates

SECONDARY OUTCOMES:
Evaluate Wound healing by wound closure | 12 weeks
  Proportion of wounds healed at 12 weeks
Evaluate wound healing by surface area reduction of greater than 40% | 4 weeks
  Proportion of wounds with surface area reduction of greater than 40% at 4 weeks
Occurrence of adverse events through case report forms | 12 weeks
  Incidence of adverse events

OTHER OUTCOMES:
Bacterial burden measured by Imaging | 12 weeks
  The effect of HaM on bacterial burden as measured by fluorescence imaging using the MolecuLight device

IPD SHARING:
Plan to Share IPD: No